CLINICAL TRIAL: NCT07216703
Title: A Phase 3, Randomized, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Sacituzumab Tirumotecan (MK-2870) in Combination With Pembrolizumab With or Without Bevacizumab Compared With Standard of Care as Firstline Maintenance Treatment for Participants With Persistent, Recurrent, or Newly Diagnosed Metastatic Cervical Cancer With PD-L1 CPS Greater Than or Equal to 1 (TroFuse-036/GOG-3123/ENGOT-cx22)
Brief Title: A Clinical Study of Sacituzumab Tirumotecan (MK-2870) in Combination With Pembrolizumab (MK-3475) as First-line Maintenance Treatment of Cervical Cancer (MK-2870-036/TroFuse-036/GOG-3123/ENGOT-cx22)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-036; U1111-1319-9926 (Registry Identifier: UTN); 2025-521514-26-00 (Registry Identifier: EU CT); MK-2870-036 (Other: MSD); TroFuse-036 (Other: MSD); GOG-3123 (Other: Gynecologic Oncology Group); ENGOT-cx22 (Other: European Network for Gynaecological Oncological Trial groups); jRCT2031250604 (Registry Identifier: jRCT (Japan Registry of Clinical Trials))
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Trophoblast Cell Surface Antigen 2 (TROP2)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Bevacizumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Participants in Part 1 Safety Run-in are allocated to a single treatment arm. Participants in study Part 2 complete induction treatment and are then randomized to 1 of 2 maintenance treatment arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Safety Run-in: Sac-TMT + Pembrolizumab + Bevacizumab (Experimental): Participants will receive sac-TMT 4 mg/kg every 2 weeks (q2w) and pembrolizumab 400 mg every 6 weeks (q6w) for up to 14 cycles (up to approximately 19 months). Bevacizumab 15 mg/kg every 3 weeks (q3w) will be administered until a treatment discontinuation criterion is met. Each cycle will be 6 weeks long.
  Interventions: Biological: Pembrolizumab; Biological: Sacituzumab Tirumotecan; Biological: Bevacizumab; Drug: Rescue Medications
- Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab (Experimental): During induction treatment, participants will receive pembrolizumab 200 mg q3w, paclitaxel 175 mg/m^2 q3w, and cisplatin 50 mg/m^2 q3w (or carboplatin area under the curve [AUC]5 mg/mL/min q3w). Participants may also receive bevacizumab 15 mg/kg q3w at the investigator's discretion. Each cycle will be 3 weeks long and treatment will continue for up to 6 cycles (up to approximately 4 months).
  During maintenance treatment, participants will receive sac-TMT 4 mg/kg q2w and pembrolizumab 400 mg q6w for up to 14 cycles (up to approximately 19 months). Participants may also receive bevacizumab 15 mg/kg q3w, at the investigator's discretion, until a treatment discontinuation criterion is met. Each cycle will be 6 weeks long.
  Interventions: Biological: Pembrolizumab; Biological: Sacituzumab Tirumotecan; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Rescue Medications
- Part 2: Pembrolizumab +/- Bevacizumab (Active Comparator): During induction treatment, participants will receive pembrolizumab 200 mg q3w, paclitaxel 175 mg/m^2 q3w, and cisplatin 50 mg/m^2 q3w (or carboplatin AUC5 mg/mL/min q3w). Participants may also receive bevacizumab 15 mg/kg q3w at the investigator's discretion. Each cycle will be 3 weeks long and treatment will continue for up to 6 cycles (up to approximately 4 months).
  During maintenance treatment, participants will receive pembrolizumab 400 mg q6w for up to 14 cycles (up to approximately 19 months). Participants may also receive bevacizumab 15 mg/kg q3w, at the investigator's discretion, until a treatment discontinuation criterion is met. Each cycle will be 6 weeks long.
  Interventions: Biological: Pembrolizumab; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) Infusion
  Other Names: Keytruda®; MK-3475; SCH 900475
Biological: Sacituzumab Tirumotecan — IV Infusion
  Other Names: sac-TMT; MK-2870; SKB264
  Arms: Part 1 Safety Run-in: Sac-TMT + Pembrolizumab + Bevacizumab; Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab
Biological: Bevacizumab — IV Infusion
  Other Names: Avastin®; Altuzan®; MVASI®
Drug: Paclitaxel — IV Infusion
  Other Names: Taxol; Onxol
  Arms: Part 2: Pembrolizumab +/- Bevacizumab; Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab
Drug: Cisplatin — IV Infusion
  Other Names: Platinol®
  Arms: Part 2: Pembrolizumab +/- Bevacizumab; Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab
Drug: Carboplatin — IV Infusion
  Other Names: Paraplatin®
  Arms: Part 2: Pembrolizumab +/- Bevacizumab; Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab
Drug: Rescue Medications — Participants receive the following rescue medications prior to sac-TMT infusion, per approved product label: histamine-1 receptor antagonist, histamine-2 receptor antagonist, acetaminophen or equivalent, and dexamethasone or equivalent. Participants are also recommended to receive prophylactic steroid mouthwash (dexamethasone or equivalent).
  Arms: Part 1 Safety Run-in: Sac-TMT + Pembrolizumab + Bevacizumab; Part 2: Sac-TMT + Pembrolizumab +/- Bevacizumab

SUMMARY:
Researchers are looking for new ways to treat metastatic cervical cancer. Cervical cancer is cancer in the cervix, the lower part of the uterus (womb). Metastatic means the cancer has spread to other parts of the body.

Researchers want to learn about giving the study medicine sacituzumab tirumotecan (also called sac-TMT or MK-2870) along with pembrolizumab and bevacizumab treatments. Sac-TMT is an antibody drug conjugate, which is a type of medicine that attaches to specific targets on cancer cells and delivers treatment to destroy those cells.

The goals of this study are to learn:

* About the safety of sac-TMT with pembrolizumab and bevacizumab, and if people tolerate them when given together, and
* If people who receive sac-TMT and pembrolizumab, with or without bevacizumab, live longer overall or without their cancer getting worse as compared to those who receive standard treatment

DETAILED DESCRIPTION:
This is a 2-part study.

In Part 1 Safety Run-in, eligible participants will be allocated to treatment with sac-TMT + pembrolizumab + bevacizumab.

In Part 2, all participants receive standard of care induction treatment. Eligible participants whose cancer does not progress then begin maintenance treatment and are randomized to receive pembrolizumab or sac-TMT + pembrolizumab. All participants in Part 2 maintenance treatment may also receive bevacizumab at the investigator's discretion.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Has a histologically confirmed diagnosis of squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of cervix
* Has persistent, recurrent, or newly diagnosed metastatic cervical cancer that is not amenable to curative treatment (surgery and/or radiation)
* If infected with human immunodeficiency virus (HIV), has well controlled HIV on antiretroviral therapy
* If positive for hepatitis B surface antigen, has received hepatitis B virus (HBV) antiviral therapy and has undetectable HBV viral load
* If has a history of hepatitis C virus (HCV) infection, has undetectable HCV viral load
* Has an Eastern Cooperative Oncology Group performance status of 0 or 1
* Has tumor programmed cell death ligand 1 expression of combined positive score ≥1

The main exclusion criteria include but are not limited to the following:

* Has HIV infection with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has received prior systemic anticancer therapy other than what is specified in this protocol
* Is currently receiving a strong inducer/inhibitor of cytochrome P450 3A4 that cannot be discontinued for the duration of treatment with sac-TMT
* Has a diagnosis of immunodeficiency
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years; replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid) is allowed
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a history of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1023 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2031-10-29 (Estimated); Study Completion 2031-10-29 (Estimated)

PRIMARY OUTCOMES:
Part 1 Safety Run-in: Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 71 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 1 Safety Run-in: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 68 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 2 Maintenance Treatment: Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 48 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first, as assessed by RECIST 1.1 as evaluated by BICR. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Part 2 Maintenance Treatment: Overall Survival (OS) | Up to approximately 60 months
  OS is defined as time from randomization to death due to any cause. OS will be presented.

SECONDARY OUTCOMES:
Part 2 Maintenance Treatment: Progression-free Survival 2 (PFS2) as Assessed by the Investigator | Up to approximately 60 months
  PFS2 is defined as the time from randomization to the documented subsequent objective disease progression after initiation of new anticancer therapy or death due to any cause, whichever occurs first. PFS2 as assessed by the investigator will be presented.
Part 2 Maintenance Treatment: Number of Participants Who Experience One or More AEs | Up to approximately 64 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 2 Maintenance Treatment: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 61 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 2 Maintenance Treatment: Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status and Quality of Life Combined Score | Baseline and up to approximately 58 months
  EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1 = Very poor to 7 = Excellent). The combined score of GHS and QoL is computed by averaging the raw scores of the 2 questions and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. A higher score indicates a better outcome. The change from baseline in the EORTC QLQ-C30 GHS and QoL combined score will be presented.
Part 2 Maintenance Treatment: Change from Baseline in EORTC QLQ-C30 Physical Functioning Combined Score | Baseline and up to approximately 58 months
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1 = Not at All to 4 = Very Much). The combined score is computed by averaging the raw scores of the 5 questions and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. A higher score indicates a better outcome. The change from baseline in the EORTC QLQ-C30 physical functioning combined score will be presented.
Part 2 Maintenance Treatment: Change from Baseline in EORTC QLQ-C30 Role Functioning Combined Score | Baseline and up to approximately 58 months
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1 = Not at All to 4 = Very Much). The combined score is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined score ranges from 0 to 100. A higher score indicates a better outcome. The change from baseline in the EORTC QLQ-C30 role functioning combined score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (3):
  - Mount Sinai Comprehensive Cancer Center ( Site 6000), Miami Beach, Florida
  - TRIALS 365 ( Site 6008), Shreveport, Louisiana
  - Women's Cancer Center of Nevada ( Site 6011), Las Vegas, Nevada
- UZ Leuven ( Site 0401), Leuven, Vlaams-Brabant, Belgium
- Nemocnice AGEL Novy Jicin a.s. ( Site 1004), Nový Jičín, Moravskoslezský kraj, Czechia
- Israel (5):
  - Hillel Yaffe Medical Center ( Site 1903), Hadera
  - Rambam Health Care Campus ( Site 1907), Haifa
  - Shaare Zedek Medical Center ( Site 1905), Jerusalem
  - Rabin Medical Center ( Site 1904), Petah Tikva
  - Sourasky Medical Center ( Site 1902), Tel Aviv
- Japan (5):
  - National Hospital Organization Hokkaido Cancer Center ( Site 2108), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 2118), Akashi, Hyōgo
  - Iwate Medical University Hospital ( Site 2116), Shiwa-gun, Iwate
  - Saitama Medical University International Medical Center ( Site 2106), Hidaka, Saitama
  - Niigata Cancer Center Hospital ( Site 2110), Niigata
- Poland (2):
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-III Klinika Radioterapii i Chemioterapii ( Site 2604), Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii. ( Site 2602), Kielce, Świętokrzyskie Voivodeship
- South Korea (5):
  - National Cancer Center ( Site 2905), Goyang-si, Kyonggi-do
  - Seoul National University Hospital ( Site 2901), Jongno-gu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 2902), Seodaemun-Gu, Seoul
  - Asan Medical Center ( Site 2904), Seoul
  - Samsung Medical Center ( Site 2903), Seoul
- National Cheng Kung University Hospital ( Site 3308), Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/